CLINICAL TRIAL: NCT07059598
Title: Evaluate the Relationship of Nutritional Status to Chemotherapy Treatment Completion Rates and Outcomes in Real-life Conditions in Patients With Metastatic and Non-metastatic Gastric, Colon, and Lung Cancer.
Brief Title: Relationship of Nutritional Status to Chemotherapy Treatment Completion and Outcomes in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA28
Record Dates: First submitted 2025-07-08; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cancer-related Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional, prospective, non-drug observational study is designed to observe the effect of the nutritional status of metastatic and non-metastatic gastric, colon and lung cancer patients on their cancer chemotherapy treatment completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Subject or subject's legally acceptable representative (LAR) has voluntarily signed and dated an ICF approved by an IEC, or any other applicable privacy authorization prior to any participation in the study.
* Ambulatory and inpatient subject.
* Subject recently (within the last month) or newly diagnosed to have metastatic or non-metastatic gastric, colon and lung cancer.
* Subject is recently receiving chemotherapy or recently prescribed to begin chemotherapy treatment per standard of care (within the last month) or candidates who will receive chemotherapy.
* Subject has a life expectancy greater than 6 months.

Exclusion Criteria:

* Subject has known dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, any other psychological condition, serious illness or medical condition that may interfere with study completion.
* Subject has malignant tumors other than treated DCIS, fully treated non-melanoma skin cancer, curatively resected in-situ cervical cancer or other curative treated tumors (except stomach, colon and lung cancer) for > 5 years.
* Subject has bone marrow metastasis.
* Subject is lactating.
* Subject is participating in another study that has not been approved as a concomitant study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Oncology Clinics
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
RMAPP | Baseline to week 24
  A tool to screen patients for risk of malnutrition and/or sarcopenia
PG-SGA | Baseline to week 24
  Healthcare Professional completed assessment resulting in score where A = Well Nourished, B = Moderately Malnourished, and C = Severely Malnourished

SECONDARY OUTCOMES:
Weight | Baseline to 24 weeks
  Change in weight
Height | Baseline
  Height in CM
Calf Circumference | Baseline to 24 weeks
  Change in calf circumference
Fat Free Mass Index | Baseline to week 24
  Evaluate Muscle Mass in relation to height and weight
EORTC QLQ-C30 | Baseline to 12 months
  Questionnaire with 28 questions from 1 to 4 with higher number is more favorable and 2 overall score questions from very poor to excellent
Body Mass Index | Baseline to week 24
  As calculated from height and weight
Handgrip Strength | Baseline to 24 weeks
  Change in handgrip dynamometer as measured in kilograms
Walking Speed | Baseline to 24 weeks
  Change in Gait Speed over 6 meter walk

OTHER OUTCOMES:
HealthCare Resource Utilization | Baseline to 12 months
  Number of unplanned inpatient hospitalizations, outpatient clinic visits, emergency department visits

CONTACTS AND LOCATIONS:
Locations (13):
- Turkey (Türkiye) (13):
  - Çukurova Üniversitesi Balcalı Hastanesi Sağlık Uygulama ve Araştırma Hastanesi, Sarıçam, Adana
  - Hacettepe Üniversitesi Tıp Fakültesi Onkoloji Hastanesi, Altındağ, Ankara
  - Ankara Etlik Şehir Hastanesi, Yenimahalle, Ankara
  - Sağlık Bilimleri Üniversitesi Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eğitim Ve Araştırma Hastanesi, Yenimahalle, Ankara
  - Bursa Uludağ Üniversitesi Tıp Fakültesi Hastanesi Sağlık Uygulama ve Araştırma Hastanesi, Ortahisar, Bursa
  - Dicle Ünversitesi Hastaneleri Tıp Fakültesi Hastanesi, Sur, Diyarbakır
  - S.B. İstanbul Medeniyet Üniversitesi Göztepe Eğitim Ve Araştırma Hastanesi, Kadıköy, Istanbul
  - İstanbul Maslak Acıbadem Hastanesi, Sarıyer, Istanbul
  - Amerikan Hastanesi, Şişli, Istanbul
  - Ege Üniversitesi Hastanesi Sağlık Uygulama ve Araştırma Merkezi, Bornova, İzmir
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Battalgazi, Malatya
  - Karadeniz Teknik Üniversitesi Farabi Hastanesi, Ortahisar, Trabzon
  - Akdeniz Üniversitesi Sağlık Araştırma ve Uygulama Merkezi Hastanesi, Antalya

IPD SHARING:
Plan to Share IPD: No